CLINICAL TRIAL: NCT00248560
Title: Phase II Study of Gemcitabine and Docetaxel (GEMDOC) Combination in Patients With Previously Treated Recurrent or Metatstatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Gemcitabine and Docetaxel in Treating Patients With Persistent, Recurrent, or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ammar Sukari, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445589; P30CA022453 (NIH); WSU-D-2830; WSU-HIC-120904M1F
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, docetaxel (Experimental): Gemcitabine given 3000 mg/m2 IV over 30 minutes and Docetaxel given 60mg/m2 IV over 60 minutes. The Docetaxel should be administered after the Gemcitabine.
  Interventions: Drug: docetaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: docetaxel — Gemcitabine given 3000 mg/m2 IV over 30 minutes and Docetaxel given 60mg/m2 IV over 60 minutes. The Docetaxel should be administered after the Gemcitabine.
  Other Names: Taxotere
Drug: Gemcitabine — Gemcitabine given 3000 mg/m2 IV over 30 minutes and Docetaxel given 60mg/m2 IV over 60 minutes. The Docetaxel should be administered after the Gemcitabine.
  Other Names: Gemzar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with docetaxel works in treating patients with persistent, recurrent, or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with previously treated persistent, recurrent, or metastatic squamous cell carcinoma of the head and neck treated with gemcitabine and docetaxel.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the duration of response and survival of patients treated with this regimen.

OUTLINE: Patients receive gemcitabine IV over 30 minutes and docetaxel IV over 60 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 4 additional courses of therapy beyond documentation of CR.

After completion of study treatment, patients are followed for survival.

PROJECTED ACCRUAL: A total of 17-41 patients will be accrued within 42-49 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck
* Metastatic, persistent, or recurrent disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Must have had definitive surgery and/or radiation therapy AND received at least 1, but no more than 2, chemotherapy regimens, either given as primary therapy or adjuvant therapy before or after surgery and/or radiotherapy
* No active or prior CNS metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* SWOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Granulocyte count > 1,500/mm^3
* Hemoglobin ≥ 8 g/dL
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin normal
* Meets 1 of the following criteria:

  * Alkaline phosphatase (AP) normal AND AST or ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST or ALT normal

Renal

* Creatinine < 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No peripheral neuropathy ≥ grade 2
* No active infection requiring systemic therapy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or any other site
* No history of severe hypersensitivity reaction to study drugs or other drugs formulated with polysorbate 80
* No other serious condition that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior taxane or gemcitabine
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered

Surgery

* See Disease Characteristics

Other

* No other concurrent therapy for this disease

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ammar Sukari, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine, Docetaxel
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Docetaxel
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Response (Complete Response [CR] + Partial Response [PR])
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: every 8 weeks for approximately 8 - 48 weeks
Measure: Number; unit: participants
Arm/Group | Gemcitabine, Docetaxel
Number analyzed (Participants) | 36
participants | 6
Statistical Analysis 1: Comparison: Gemcitabine, Docetaxel; Test type: Superiority or Other; Response rate = 0.17, 95% CI 2-sided [0.08 to 0.32]

2. Secondary Outcome: Response Duration
Description: Response duration in months
Time Frame: Every 8 weeks
Population: Only those patients that have a recorded CR or PR
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Docetaxel
Number analyzed (Participants) | 6
months | 3.2 [2.0 to 6.1]

3. Secondary Outcome: Survival
Description: Overall Survival using the Kaplan-Meier method
Time Frame: Every 8 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Docetaxel
Number analyzed (Participants) | 36
months | 4.2 [2.4 to 7.0]

4. Secondary Outcome: Toxicity as Measured by Number and Grade of Adverse Events
Description: Toxicity as the total number of participants with a given grade 3 and/or grade 4 adverse event
Time Frame: Every 2 weeks
Measure: Number; unit: participants
Arm/Group | Gemcitabine, Docetaxel
Number analyzed (Participants) | 36
participants
  Anemia | 13
  Neutropenia | 10
  Hyponatremia | 10
  Dehydration | 3
  Fatigue | 3
  Dyspnea | 3
  Pneumonia | 3
  Thrombocytopenia | 2
  Febrile neutropenia | 1
  Tachycardia | 1
  Syncope | 1
  Fluid retention | 1
  Mucositis | 1
  Hyperglycemia | 1
  Constipation | 1
  Anorexia | 1
  Vomiting | 1
  Other non-hematologic toxicity | 1

ADVERSE EVENTS:
Arm/Group | Gemcitabine, Docetaxel
Serious Adverse Events (participants affected / at risk) | 25/36
Other Adverse Events (participants affected / at risk) | 33/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Docetaxel (N=36)
Anemia (Blood and lymphatic system disorders) | 13 (13)
Neutropenia (Blood and lymphatic system disorders) | 10 (10)
Hyponatremia (Metabolism and nutrition disorders) | 10 (10)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Fluid Retention (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Gemcitabine, Docetaxel (N=36)
Nausea (Gastrointestinal disorders) | 3/28 (6)
Anemia (Blood and lymphatic system disorders) | 19 (19)
Neutropenia (Blood and lymphatic system disorders) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Fatigue (General disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (15)
Tachycardia (Cardiac disorders) | 4 (4)
Fluid Retention (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5)
Creatinine (Investigations) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
The trial design was changed during accrual to allow for study continuation although response rate was lower than predicted. The trial was completed but it did not meet the specified end points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No